CLINICAL TRIAL: NCT07003295
Title: A Phase II Study of Glofitamab for Relapsed/Refractory Mantle Cell Lymphoma in Patients Previously Treated With CD19-Directed CAR T-Cell Therapy
Brief Title: Testing the Anti-cancer Drug, Glofitamab, in Patients With Mantle Cell Lymphoma (A Type of Blood Cancer) Whose Disease Returned After CAR-T Cell Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2025-03915; NCI-2025-03915 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10702 (Other: JHU Sidney Kimmel Comprehensive Cancer Center LAO); 10702 (Other: CTEP); UM1CA186691 (NIH)
Record Dates: First submitted 2025-06-03; First posted 2025-06-04 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Recurrent Mantle Cell Lymphoma; Refractory Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Specimen Handling; glofitamab; obinutuzumab; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (obinutuzumab, glofitamab) (Experimental): Patients receive obinutuzumab IV on day 1 or on days 1 and 2 of cycle 1 and glofitamab IV over 8 hours on days 8 and 15 of cycle 1 then over 2-8 hours on day 1 of cycles 2-12. Cycles repeat every 21 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection and PET/CT throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Glofitamab; Biological: Obinutuzumab; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Biological: Glofitamab — Given IV
  Other Names: Anti-CD20 x Anti-CD3 Bispecific Monoclonal Antibody RO7082859; Columvi; Glofitamab-gxbm; RO 7082859; RO-7082859; RO7082859
Biological: Obinutuzumab — Given IV
  Other Names: Anti-CD20 Monoclonal Antibody R7159; GA 101; GA-101; GA101; Gazyva; huMAB(CD20); R 7159; R-7159; R7159; RO 5072759; RO-5072759; RO5072759
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT

SUMMARY:
This phase II trial tests the safety and side effects of glofitamab and obinutuzumab and how well they work in treating patients with mantle cell lymphoma that has come back after a period of improvement (relapsed) or that has not responded to previous treatment (refractory) after receiving CD19-directed chimeric antigen receptor (CAR) T-cell therapy. CAR T-cell therapy is a form of immunotherapy where the immune system cell, T-cell, is changed to attack cancer cells. Glofitamab is a bispecific antibody that can bind to two different antigens at the same time. Glofitamab binds to CD3, a protein found on T cells (a type of white blood cell), and CD20 a protein found on B cells (another type of white blood cell) and some lymphoma cells. This may help the immune system kill cancer cells. Obinutuzumab is a monoclonal antibody that may interfere with the ability of cancer cells to grow and spread. A monoclonal antibody is a type of protein that can bind to certain targets in the body, such as molecules that cause the body to make an immune response (antigens). Giving glofitamab and obinutuzumab may be safe, tolerable, and/or effective in treating patients with relapsed or refractory mantle cell lymphoma after receiving CD19-directed CAR T-cell therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the proportion of relapsed/refractory (R/R) mantle cell lymphoma (MCL) patients with an objective response (OR) to glofitamab after prior treatment with chimeric antigen receptor (CAR)-T.

SECONDARY OBJECTIVES:

I. To describe the proportion of patients with a complete response (CR). II. To describe the progression-free survival (PFS) and overall survival (OS) at 24 months.

III. To describe the incidence of grade 3-4 cytokine release syndrome (CRS). IV. To describe the incidence of grade 3-4 neurologic toxicity. V. To describe the relationship between glofitamab clearance at baseline, changes in clearance over time, treatment response, and duration of response.

EXPLORATORY OBJECTIVES:

I. To evaluate the relationship between circulating tumor deoxyribonucleic acid (DNA) (ctDNA) detection in plasma, treatment response, and duration of response.

II. To evaluate the relationship between CAR T-cell levels in plasma, immunophenotype, treatment response, and duration of response.

III. To evaluate the relationship between fluorodeoxyglucose positron emission tomography/ computed tomography (FDG PET/CT) interlesional treatment response heterogeneity and survival outcomes.

IV. To evaluate the relationship between organ-specific changes in standardized uptake value (SUV) metrics and immune-related adverse events (AEs).

OUTLINE:

Patients receive obinutuzumab intravenously (IV) on day 1 or on days 1 and 2 of cycle 1 and glofitamab IV over 8 hours on days 8 and 15 of cycle 1 then over 2-8 hours on day 1 of cycles 2-12. Cycles repeat every 21 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection and PET/CT throughout the study.

After completion of study treatment, patients are followed every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed diagnosis of mantle cell lymphoma that is relapsed (disease progression after the last treatment regimen) or refractory (failure to achieve a partial or complete response from the last treatment regimen)
* Patients must have been previously treated with an anti-CD19 CAR T-cell therapy and have failed or been intolerant to Bruton's tyrosine kinase (BTK) inhibition. Both commercial and investigational CAR-T products which target CD19 will be allowed, including dual-targeting products
* Patients must have at least one bi-dimensionally measurable (defined as at least 1.5 cm) nodal lesion or one bi-dimensionally measurable (at least 1 cm) extranodal lesion, as measured on CT scan
* Age ≥ 18 years. Because no dosing or adverse event (AE) data are currently available on the use of glofitamab and obinutuzumab in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 60%)
* Absolute neutrophil count ≥ 1,000/mcL
* Platelets ≥ 50,000/mcL
* Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) or ≤ 3 x institutional ULN if the patient has Gilbert syndrome
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamic pyruvic transaminase [SGPT]) ≤ 3 x institutional ULN
* Creatinine ≤ 1.5 x institutional ULN OR glomerular filtration rate (GFR) ≥ 60 mL/min/1.73 m^2
* Patients with human immunodeficiency virus (HIV) infection are eligible if on effective anti-retroviral therapy with undetectable viral load within 6 months
* Patients with a history of hepatitis B virus (HBV) infection or positive total hepatitis B core antibody (HBcAb) are eligible if the hepatitis B surface antigen (HBsAg) is negative and HBV DNA viral load is undetectable by polymerase chain reaction (PCR) at the time of screening. Such patients must be managed with appropriate anti-viral therapy, if indicated, and must be willing to undergo HBV DNA testing on day 1 of each cycle and every 3 months for at least 12 months after the final cycle of study treatment
* Patients with a history of hepatitis C virus (HCV) infection or positive HCV antibody are eligible if HCV ribonucleic acid (RNA) viral load is undetectable by PCR
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression and patients are asymptomatic from CNS involvement
* Patients with new, progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that patients are asymptomatic and immediate CNS specific treatment is not required and is unlikely to be required during the first cycle of therapy
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial, such as patients with prostate cancer or breast cancer receiving hormonal therapy
* The effects of glofitamab and obinutuzumab on the developing human fetus are unknown. For this reason and because glofitamab and obinutuzumab are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 2 months after completion of glofitamab and 6 months after completion of obinutuzumab administration. Women of childbearing potential must use effective contraceptive precautions 2 months after completion of glofitamab treatment and 18 months after the last dose of obinutuzumab treatment
* Ability to understand and the willingness to sign a written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants

Exclusion Criteria:

* Patients who have not recovered from AEs due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia
* Patients who are receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to glofitamab and obinutuzumab
* Pregnant women are excluded from this study because glofitamab and obinutuzumab are agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for AEs in nursing infants secondary to treatment of the mother with glofitamab and obinutuzumab, breastfeeding should be discontinued if the mother is treated with glofitamab and obinutuzumab
* Patients with active CRS or requiring intervention for CRS within 14 days prior to study enrollment
* Patients with active neurotoxicity or requiring intervention for neurotoxicity within 14 days prior to study enrollment
* Patients requiring antimicrobial treatment or hospitalization for active infection within 14 days prior to study enrollment for known active bacterial, viral (including severe acute respiratory syndrome coronavirus 2 [SARS-CoV-2]), fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds). Infection must be completely resolved prior to initiation of study treatment
* Patients receiving systemic immunosuppressive medications within 14 days prior to study enrollment, including, but not limited to: prednisone ≥ 20 mg per day, azathioprine, methotrexate, anti-tumor necrosis factor agents, anti-interleukin-6/6R agents, or anti-interleukin 1 agents, are not eligible. The use of inhaled corticosteroids is permitted
* Patients with known or suspected chronic active Epstein Barr virus (EBV) or cytomegalovirus (CMV) infection
* Patients with known or suspected history of hemophagocytic lymphohistiocytosis (HLH)
* Patients with prior treatment with glofitamab or other bispecific antibodies targeting both CD20 and CD3
* Patients with known history of progressive multifocal leukoencephalopathy
* Patients with current or past history of CNS disease, such as stroke, epilepsy, CNS vasculitis, or neurodegenerative disease. Patients with a history of stroke who have not experienced a stroke or transient ischemic attack in the past 2 years and have no residual neurologic deficits as judged by the investigator are allowed
* Patients with the significant cardiovascular disease, including New York Heart Association class III or IV or otherwise symptomatic heart failure (stage C or D), myocardial infarction within the last 3 months, unstable arrhythmias, or unstable angina
* Patients who have undergone major surgery for non-diagnostic purposes within 4 weeks before first study treatment
* Patients who have received a live attenuated vaccine within 4 weeks before first study treatment administration or anticipation that such a live, attenuated vaccine will be required during the study
* Patients with a positive SARS-CoV-2 test 7 days prior to enrollment
* Patients with current or past history of Waldenström macroglobulinemia
* Patients with an active autoimmune disease that could be exacerbated by immunotherapy, excluding those with a remote history or well-controlled autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-08-14 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Up to 2 years
  A Simon 2-stage optimal design will be used with a favorable response of 55% and unfavorable response of 25%.

SECONDARY OUTCOMES:
Complete response rate | Up to 2 years
  Proportions will be estimated with Agresti-Coull 95% binomial confidence intervals.
Progression-free survival (PFS) | Up to 24 months
  Proportions will be estimated with Agresti-Coull 95% binomial confidence intervals. Will be estimated using the Kaplan Meier method. Estimates of PFS will be reported with a 95% confidence interval.
Overall survival (OS) | Up to 24 months
  Proportions will be estimated with Agresti-Coull 95% binomial confidence intervals. Will be estimated using the Kaplan Meier method. Estimates of OS will be reported with a 95% confidence interval.
Incidence of grade 3-4 cytokine release syndrome | Up to 2 years
  Proportions will be estimated with Agresti-Coull 95% binomial confidence intervals. Incidence will be described.
Incidence of grade 3-4 neurologic toxicity | Up to 2 years
  Proportions will be estimated with Agresti-Coull 95% binomial confidence intervals. Incidence will be described.
Changes in glofitamab clearance | At baseline and up to 2 years
  Pharmacokinetics (PK) of glofitamab will also be determined to assess exposure-response and clearance-response relationships. When appropriate, Bayesian logistic regression analysis will be performed to assess exposure-response and clearance-response relationships. Basic non-compartmental analyses will be performed with the concentration versus time data to summarize several pharmacokinetic parameters including observed maximum concentration and area under the observed concentration versus time curves. Descriptive statistics will be used to summarize these results. Nonlinear mixed-effects modeling will also be performed to develop a population PK model of glofitamab to describe PK properties, including absorption, distribution, and overall elimination.

OTHER OUTCOMES:
Relationship in circulating tumor deoxyribonucleic acid (ctDNA) in plasma, treatment response, and duration of response | On day 1 of cycles 1, 3, and 5 (cycle length = 21 days)
  Descriptive statistics will be used to summarize the ctDNA results.
Relationship between chimeric antigen receptor (CAR) T-cell levels in plasma, immunophenotype, treatment response, and duration of response | On day 1 of cycles 1, 3 and 5 (cycle length = 21 days)
  Descriptive statistics will be used to summarize the CAR-T and T-cell immunophenotype results.
Glofitamab PK | Before and 5-60 minutes after glofitamab infusions on day 8 of cycle 1 and day 1 of cycles 2-4, 6, 9, and 12 (cycle length = 21 days)
Relationship between fluorodeoxyglucose positron emission tomography/ computed tomography interlesional treatment response heterogeneity and survival outcomes | At baseline and after cycles 2, 5, 8, and 12 (cycle length = 21 days)
  Responses will be assessed using 2014 revised response criteria as outlined by Cheson et al., 2014.
Relationship between organ-specific changes in standardized uptake value (SUV) metrics and immune-related adverse events (AEs) | At baseline and after cycles 2, 5, 8, and 12 (cycle length = 21 days)
  Images will be analyzed for changes in SUV metrics using the TRAQinform tool. Changes in SUV metrics (including max, mean, total) will be obtained in each lesion with metrics reported numerically, as well as graphically to understand treatment response heterogeneity (percent lesions for each response classification based on each SUV metric and change in lesion based on established limits of agreement). The automated organ segmentations will be used to quantify organ uptake, which will be correlated with occurrence of AEs in those organs. A TRAQinform profile based on an artificial intelligence model (random survival forest model generated in lymphoma) of survival will be used to explore predictive accuracy in patients treated with glofitamab.

CONTACTS AND LOCATIONS:
Overall Officials: Cole H Sterling, Principal Investigator — JHU Sidney Kimmel Comprehensive Cancer Center LAO
Locations (1):
- JHU Sidney Kimmel Comprehensive Cancer Center LAO, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm